CLINICAL TRIAL: NCT01877720
Title: Physiologic Comparison Between Noninvasive Neurally Adjusted Ventilatory Assist (NAVA) and Pressure Support (PS) in Preterm Infants
Brief Title: Physiologic Comparison Between NIV-NAVA and PS in Preterm Infants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Rotary (Unknown)
Responsible Party: Principal Investigator, Han-Suk Kim, MD, PhD, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NIV-NAVA Physiologic Study
Record Dates: First submitted 2013-06-05; First posted 2013-06-14 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-11

CONDITIONS: Noninvasive Neurally Adjusted Ventilatory Assist and Pressure Support in Preterm Infants
Keywords: Preterm infant less than 32 weeks of gestation age; intubated more than 48 hours after birth; postextubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAVA-PS (Experimental): noninvasive NAVA first for 15 minutes and then PSV for 15 minutes
  Interventions: Device: noninvasive respiratory support with NAVA mode and PSV
- PS-NAVA (Experimental): noninvasive PSV first for 15 minutes and then NAVA for 15 minutes
  Interventions: Device: noninvasive respiratory support with NAVA mode and PSV

INTERVENTIONS:
Device: noninvasive respiratory support with NAVA mode and PSV

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) has been shown to improve patient- ventilator interaction and reduce asynchronies. This is a short-term physiologic comparison between PSV (pressure support ventilation) and NAVA in delivering noninvasive ventilation through a nasal cannula, in premature infants postextubation. Patients will undergo a 30-min crossover trial of noninvasive PSV and NAVA, 15 minutes each. Diaphragm electrical activity (EAdi)and airway pressure (Paw) are recorded to derive neural and mechanical respiratory rate and timing, inspiratory trigger delays time of synchrony between diaphragm contraction and ventilator assistance, and the asynchrony index (AI).

ELIGIBILITY:
Inclusion Criteria:

* preterm infants less than 32 weeks of gestational age
* intubated more than 48 hours after birth
* subjected to extubation with minimal ventilator setting (mean airway pressure < 7cmH2O + peak inspiratory pressure < 13 cmH2O + FiO2 < 0.4 + respiratory rate < 35/min)
* with informed consent from parents

Exclusion Criteria:

* with major congenital anomalies
* use of sedative or anesthetic drugs
* hemodynamic instability
* grade 3 or higher intraventricular hemorrhage
* phrenic nerve palsy

Ages: 3 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han-Suk Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Bundang, Gyeonggi-do
  - Seoul National University Children's Hospital, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Lee J, Kim HS, Jung YH, Shin SH, Choi CW, Kim EK, Kim BI, Choi JH. Non-invasive neurally adjusted ventilatory assist in preterm infants: a randomised phase II crossover trial. Arch Dis Child Fetal Neonatal Ed. 2015 Nov;100(6):F507-13. doi: 10.1136/archdischild-2014-308057. Epub 2015 Jul 15. PMID 26178463

RESULTS

PARTICIPANT FLOW:
Groups:
- PS-NAVA: noninvasive PSV first for 15 minutes and then NAVA for 15 minutes
  crossover of noninvasive respiratory support with NAVA mode and PSV
- NAVA-PS: noninvasive NAVA first for 15 minutes and then PSV for 15 minutes
  crossover of noninvasive respiratory support with NAVA mode and PSV
Period: Overall Study
Arm/Group | PS-NAVA | NAVA-PS
Started | 8 | 8
1st Intervention | 7 | 8
2nd Intervention | 7 | 8
Completed | 7 | 8
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Enrolled Patients
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: weeks of gestation]
  Gestational age | 27.1 [26.0 to 28.2]
Age, Continuous [Median (Inter-Quartile Range); unit: day]
  Postnatal age at study | 25 [17.5 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Birth weight [Median (Inter-Quartile Range); unit: g] | 790 [675 to 1215]

OUTCOME MEASURES:

1. Primary Outcome: Trigger Delay
Description: Inspiratory trigger delay could be calculated by the time interval between beginning of the increase of actual diaphragmatic excitation and start of ventilator inspiratory flow of each respiration. The value will be present as a mean of all inspiratory trigger delay measurements of all respiration during last 5 minutes of each 15 minutes trial.
Time Frame: last 5-min of each 15-min trial
Measure: Mean (Standard Deviation); unit: ms
Groups:
- NIV-NAVA: non-invasive NAVA
- NIV-PS: non-invasive PS
Arm/Group | NIV-NAVA | NIV-PS
Number analyzed (Participants) | 15 | 15
ms | 35.2 (8.3) | 294.6 (101.9)
Statistical Analysis 1: Comparison: NIV-NAVA vs NIV-PS; Test type: Superiority or Other; p < 0.001, Paired t-test

2. Secondary Outcome: Ti_excess (Inspiratory Time in Excess)
Description: Ti_excess = (VPT-NIT)/NIT
  VPT: ventilator pressurization time (VPT) between beginning and end of inspiratory flow NIT: neural inspiratory time (NIT) between beginning of the increase in the diaphragmatic excitation and its maximal value
Time Frame: last 5-min of each 15-min trial
Measure: Mean (Standard Deviation); unit: percentage of neural inspiratory time
Arm/Group | NIV-NAVA | NIV-PS
Number analyzed (Participants) | 15 | 15
percentage of neural inspiratory time | 32.2 (11.4) | 56.8 (25.2)
Statistical Analysis 1: Comparison: NIV-NAVA vs NIV-PS; Test type: Superiority or Other; p = 0.001, Paired t-test

3. Secondary Outcome: Minute Ventilation Volume
Description: inspiratory tidal volume / respiratory rate
Time Frame: last 5-min of each 15-min trial
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | NIV-NAVA | NIV-PS
Number analyzed (Participants) | 15 | 15
mL/kg/min | 114.9 (47.0) | 124.1 (42.4)
Statistical Analysis 1: Comparison: NIV-NAVA vs NIV-PS; Test type: Superiority or Other; p = 0.74, Paired t-test

4. Secondary Outcome: Peak Inspiratory Pressure
Time Frame: last 5-min of each 15-min trial
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | NIV-NAVA | NIV-PS
Number analyzed (Participants) | 15 | 15
cmH2O | 12.3 (1.5) | 14.7 (2.7)
Statistical Analysis 1: Comparison: NIV-NAVA vs NIV-PS; Test type: Superiority or Other; p = 0.003, Paired t-test

5. Secondary Outcome: Pneumatic Respiratory Rate
Time Frame: last 5-min of each 15-min trial
Measure: Mean (Standard Deviation); unit: breaths per min
Arm/Group | NIV-NAVA | NIV-PS
Number analyzed (Participants) | 15 | 15
breaths per min | 46.3 (12.6) | 33.3 (13.1)
Statistical Analysis 1: Comparison: NIV-NAVA vs NIV-PS; Test type: Superiority or Other; p = 0.002, Paired t-test

6. Secondary Outcome: Maximum EAdi
Time Frame: last 5-min of each 15-min trial
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | NIV-NAVA | NIV-PS
Number analyzed (Participants) | 15 | 15
uV | 12.6 (6.3) | 16.6 (8.7)
Statistical Analysis 1: Comparison: NIV-NAVA vs NIV-PS; Test type: Superiority or Other; p = 0.003, Paired t-test

7. Secondary Outcome: Swing EAdi
Time Frame: last 5-min of each 15-min trial
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | NIV-NAVA | NIV-PS
Number analyzed (Participants) | 15 | 15
uV | 8.8 (4.8) | 12.2 (8.7)
Statistical Analysis 1: Comparison: NIV-NAVA vs NIV-PS; Test type: Superiority or Other; p = 0.012, Paired t-test

8. Secondary Outcome: Leakage
Description: [TVi (inspiratory tidal volume) - TVe (expiratory tidal volume)]/TVi (inspiratory tidal volume)
Time Frame: last 5-min of each 15-min trial
Measure: Mean (Standard Deviation); unit: percentage of inspiratory tidal volume
Arm/Group | NIV-NAVA | NIV-PS
Number analyzed (Participants) | 15 | 15
percentage of inspiratory tidal volume | 87.6 (8.3) | 86.7 (6.8)
Statistical Analysis 1: Comparison: NIV-NAVA vs NIV-PS; Test type: Superiority or Other; p = 0.67, Paired t-test

9. Secondary Outcome: All Asynchrony Events
Time Frame: last 5-min of each 15-min trial
Measure: Median (Inter-Quartile Range); unit: events per min
Arm/Group | NIV-NAVA | NIV-PS
Number analyzed (Participants) | 15 | 15
events per min | 8.2 [3.0 to 11.5] | 47.6 [38.1 to 61.1]
Statistical Analysis 1: Comparison: NIV-NAVA vs NIV-PS; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test

10. Secondary Outcome: Asynchrony Index
Description: total number of each event per minute
  1. ineffective efforts: presence of a characteristic EAdi (electrical activity of diaphragm) activity not followed by a ventilator delivered pressurization
  2. auto-triggering: a cycle delivered by the ventilator without EAdi signal
  3. premature cycling
  4. delayed cycling: VPT > NIT x2
  5. double triggering
     * Asynchrony index = [(1)+(2)+(3)+(4)+(5)]/[(1)+pneumatic respiratory rate] x100
Time Frame: last 5-min of each 15-min trial
Measure: Median (Inter-Quartile Range); unit: percentage of neural respiration
Arm/Group | NIV-NAVA | NIV-PS
Number analyzed (Participants) | 15 | 15
percentage of neural respiration | 19.7 [9.6 to 23.4] | 73.9 [71.5 to 78.1]
Statistical Analysis 1: Comparison: NIV-NAVA vs NIV-PS; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test

11. Secondary Outcome: SpO2
Description: transcutaneous peripheral saturation of oxygen by pulse oximeter
Time Frame: last 5-min of each 15-min trial
Reporting Status: Not Posted

12. Secondary Outcome: Heart Rate
Time Frame: last 5-min of each 15-min trial
Reporting Status: Not Posted

13. Secondary Outcome: Blood Pressure
Description: systolic, diastolic and mean blood pressure measured by non-invasive cuff
Time Frame: last 5-min of each 15-min trial
Reporting Status: Not Posted

14. Secondary Outcome: Respiratory Rate
Time Frame: last 5-min of each 15-min trial
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | NIV-NAVA | NIV-PS
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIV-NAVA (N=15) | NIV-PS (N=15)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — Bradycardia longer than 2 min

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No